CLINICAL TRIAL: NCT05316350
Title: Validation of HWA10 With Withings ECG-app for the Detection of Atrial Fibrillation
Brief Title: Withings ECG-app Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Withings (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HWA10-ECG
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Atrial Fibrillation
Keywords: mhealth; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Atrial Fibrillation (Experimental)
  Interventions: Device: Electrocardiogram recording
- Normal Sinus Rhythm (Experimental)
  Interventions: Device: Electrocardiogram recording

INTERVENTIONS:
Device: Electrocardiogram recording — ECG recording with investigational device
Device: Electrocardiogram recording — ECG recording with reference device

SUMMARY:
The aim of the study is to evaluate the performance of Withings HWA10 with embedded Withings ECG-app in the automatic detection of atrial fibrillation

ELIGIBILITY:
Inclusion Criteria:

* Male or female who are 22 years of age or older
* Subject able to read, understand, and provide written informed consent
* Subject willing and able to participate in the study procedures as described in the consent form
* Subject able to communicate effectively with and willing to follow instructions from the study staff
* Have a wrist circumference between 140 mm and 210 mm (measured at "band center" on the preferred wrist, 1cm from the bone. This location is determined by asking the volunteer to put on a normal wrist-watch and marking the skin with a pen/marker to outline the edges of the band.)

Exclusion Criteria:

* Vulnerable subject with regard to regulations in force

  * Subject who is deprived of liberty by judicial, medical or administrative decision,
  * Underage subject,
  * Legally protected subject, or subject who is unable, linguistic or psychic incapacity, to sign the written informed consent form,
* Subject within several of the above categories,
* Subject who refused to participate in the study,
* Subject mentally impaired resulting in limited ability to cooperate
* Subject in physical incapacity to wear a watch on one wrist and place the other hand on top of the watch
* Subject with electrical stimulation by pacemaker
* Patient with pathologic disorder that may affect motricity resulting in significant tremor that prevents subject from being able to hold still (e.g Parkinson disease)
* Acute myocardial infarction (MI) within 90 days of screening or other cardiovascular disease that, in the opinion of the Investigator, may increase the risk to the subject or renders data uninterpretable (e.g., recent or ongoing unstable angina, decompensated heart failure, active myocarditis or pericarditis)
* Acute pulmonary embolism or pulmonary infarction, within 90 days of screening
* Stroke or transient ischemic attack within 90 days of screening
* Active life-threatening rhythms as determined by the investigator (ventricular tachycardia, ventricular fibrillation, 3 rd -degree heart block).
* History of abnormal life-threatening rhythms (ventricular tachycardia, ventricular fibrillation, 3 rd -degree heart block)
* Symptomatic (or active) allergic skin reactions such as eczema, rosacea, impetigo, dermatomyositis or allergic contact dermatitis on both wrists or over electrode attachment sites
* Known sensitivity to medical adhesives, isopropyl alcohol, watch bands, or electrocardiogram (ECG) electrodes including known allergy or sensitivity to fluoroelastomer bands primarily used in wrist worn fitness devices

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 685 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Co-primary outcomes | 4 months
  Sensitivity (percentage of true positives) in detecting AF from conclusive recordings generated by the software under test, that is recordings resulting in a classification of AF or SR by the SUT, compared to the reference 12-lead ECG.
Co-primary outcomes | 4 months
  Specificity (percentage of true negatives) in detecting AF from conclusive recordings generated by the software under test, that is recordings resulting in a classification of AF or SR by the SUT, compared to the reference 12-lead ECG.

SECONDARY OUTCOMES:
Evaluation of the classification into heart rate subgroups | 4 months
  The classification into heart rate subgroups will be evaluated for the pairs of strips such that the rhythm classification of the 12-lead ECG is either SR or AF and such that the strip generated by the SUT is classified as either SR or AF. The evaluation will be assessed with the concordance of classifications, i.e. the percentage P of identical classifications by the SUT and the reference method, into each of the four following subgroups:
  * SR with a HR between 50 and 99 bpm
  * SR with a HR between 100 and 150 bpm
  * AF with a HR between 50 and 99 bpm
  * AF with a HR between 100 and 150 bpm
Clinical Equivalence of ECG waveforms | 4 months
  Clinical Equivalence of ECG waveforms will be qualitatively and quantitatively assessed between the 6-leads generated by the SUT and the leads I, II, III, aVR, aVL, aVF of the 12-lead ECG by a board of certified cardiologists:
  The visibility and polarity of the P waves, QRS complexes and T waves will be determined by cardiologists and according to a set of predetermined rules. For each type of wave (P, QRS and T),
Clinical Equivalence of ECG waveforms | 4 months
  The durations of the QT intervals, QRS complex widths, and PR intervals will be measured by cardiologists with a caliper and according to a set of predetermined rules for each of the 6 leads of the strips generated by the SUT and the leads I, II, III, aVR, aVL, aVF of the 12-lead ECG.
Heart Rate equivalence | 4 months
  heart rate will be determined by independent cardiologists, or cardiac technicians supervised by cardiologists, from each six-channel strip recorded with the SUT and from each lead I, II, III, aVR, aVL, aVF of the 12-lead reference ECG

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Wessler, MD, Principal Investigator — Heartbeat Health
Locations (10):
- United States (9):
  - FWD Clinical Research, Boca Raton, Florida
  - Florida Cardiovascular Research, Hialeah, Florida
  - Diverse Clinical Research, Miami, Florida
  - The Angel Medical Research, Miami Lakes, Florida
  - American Institute of Therapeutics, Lake Bluff, Illinois
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Heartbeat Health, New York, New York
  - Texas Heart Institute, Houston, Texas
  - LINQ Research LLC, Pearland, Texas
- Henri-Mondor Hospital, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No